CLINICAL TRIAL: NCT01345136
Title: A Single Arm, Monocenter Phase II Trial of RAD001 as Monotherapy in the Treatment of Neurofibromatosis Type 2 - Related Vestibular Schwannoma
Brief Title: Study of RAD001 for Treatment of NF2-related Vestibular Schwannoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-001492
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Neurofibromatosis Type 2; Neuroma, Acoustic
Keywords: Neurofibromatosis Type 2; Vestibular schwannoma; Hearing
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 Treatment (Experimental): All subjects will be given RAD001 for 1 year (12 months).
  Interventions: Drug: RAD001, everolimus

INTERVENTIONS:
Drug: RAD001, everolimus — Adults: 10 mg p.o. daily dose, age 16 - 17: 3.0 mg/m2 p.o. daily
  Other Names: Everolimus; Afinitor

SUMMARY:
The purpose of the study is to determine if RAD001 treatment will shrink or slow the growth of the vestibular schwannoma(s) in Neurofibromatosis 2 (NF2) patients. Secondary objectives include determining if RAD001 treatment will improve hearing ability in NF2 patients.

RAD001 is an oral drug that is approved by Food and Drug Administration (FDA) for other types of tumors, it is not approved by the FDA for treatment of NF2 related tumors.

DETAILED DESCRIPTION:
This protocol is a Phase II, open-label, efficacy and safety study of single-agent RAD001 in patients with NF2. During the study, subjects will receive continuous daily oral treatment with RAD001 for up to 1 year or until tumor progression.

Primary Objective: To determine whether RAD001 has an effect on the VS growth in patients with NF2 at a rate sufficient to submit the drug for further testing.

Secondary Objectives: To determine whether RAD001 has an effect on the volume of other intracranial tumors, and to assess the effect of RAD001 on hearing function in patients with NF2 (when applicable).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NF2 by National Institutes of Health (NIH) criteria
* Age ≥ 16 years
* Progressive VS growth during the previous 12 months.
* WHO performance status > or = 2
* Adequate bone marrow, liver and renal function.
* For women of childbearing potential, no pregnancy or breast-feeding
* Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Willingness to provide informed consent

Exclusion Criteria:

* Inability to tolerate periodic MRI scans or gadolinium contrast.
* Inability to tolerate periodic audiologic testing or to understand a language with established scoring for word recognition testing.
* Inability to adequately perform volumetric measurement of at least 1 target lesionNote: Patients with cochlear or auditory brainstem implants may participate if a target lesion can be accurately assessed.
* Radiation therapy for the target lesion in the 60 months preceding inclusion in the study.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug.
* Immunization with attenuated live vaccines within one week of study entry or during study period.
* Presence of a fungal infection requiring systemic antifungal treatment at enrollment
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions.
* Patients with a known hypersensitivity to everolimus or other types of rapamycin or to its excipients.
* Patients unwilling to or unable to comply with the protocol

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Vestibular schwannoma volume | 1 year (12 months)
  Determine the effect of RAD001 on change in vestibular schwannoma volume (mm3) by MRI from baseline to 1 year.

SECONDARY OUTCOMES:
Hearing | 1 year (12 months)
  Determine the effects of RAD001 treatment on hearing changes (from baseline to 1 year in the ear with the growing vestibular schwannoma.
Number of adverse events | 1 year, 1 month (13 months)
  Determine the number of study subjects with adverse events by grade of severity

CONTACTS AND LOCATIONS:
Overall Officials: Marco Giovannini, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Giovannini M, Bonne NX, Vitte J, Chareyre F, Tanaka K, Adams R, Fisher LM, Valeyrie-Allanore L, Wolkenstein P, Goutagny S, Kalamarides M. mTORC1 inhibition delays growth of neurofibromatosis type 2 schwannoma. Neuro Oncol. 2014 Apr;16(4):493-504. doi: 10.1093/neuonc/not242. Epub 2014 Jan 10. PMID 24414536
- [Background] Goutagny S, Raymond E, Esposito-Farese M, Trunet S, Mawrin C, Bernardeschi D, Larroque B, Sterkers O, Giovannini M, Kalamarides M. Phase II study of mTORC1 inhibition by everolimus in neurofibromatosis type 2 patients with growing vestibular schwannomas. J Neurooncol. 2015 Apr;122(2):313-20. doi: 10.1007/s11060-014-1710-0. Epub 2015 Jan 8. PMID 25567352
- [Derived] Nghiemphu PL, Vitte J, Dombi E, Nguyen T, Wagle N, Ishiyama A, Sepahdari AR, Cachia D, Widemann BC, Brackmann DE, Doherty JK, Kalamarides M, Giovannini M. Imaging as an early biomarker to predict sensitivity to everolimus for progressive NF2-related vestibular schwannoma. J Neurooncol. 2024 Apr;167(2):339-348. doi: 10.1007/s11060-024-04596-4. Epub 2024 Feb 19. PMID 38372904